CLINICAL TRIAL: NCT01315691
Title: Randomized, Placebo-Controlled, Double-Blind, Multicenter Study to Assess the Efficacy, Safety and Tolerability of Arikace™ in Cystic Fibrosis Patients With Chronic Infection Due to Pseudomonas Aeruginosa
Brief Title: Study to Evaluate Arikace™ in CF Patients With Chronic Infection Due to Pseudomonas Aeruginosa
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TR02-109
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Respiratory Infections; Pulmonary Cystic Fibrosis; Amikacin; Anti-bacterial agents
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Infections | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arikace™ (Experimental): Liposomal amikacin for inhalation
  Interventions: Drug: Liposomal amikacin for inhalation
- Placebo (Placebo Comparator): Placebo for liposomal amikacin for inhalation
  Interventions: Drug: Placebo for liposomal amikacin for inhalation

INTERVENTIONS:
Drug: Liposomal amikacin for inhalation — * Liposomal amikacin for inhalation is provided as a sterile aqueous liposomal dispersion for inhalation via nebulization.
  * 590 mg of liposomal amikacin for inhalation is administered once daily using the PARI Investigational eFlow® Nebulizer.
  * Administration time is approximately 13 minutes.
  * Liposomal amikacin for inhalation will be administered for 28 days followed by 56 days off treatment.
  Arms: Arikace™
Drug: Placebo for liposomal amikacin for inhalation — * Placebo is provided as a sterile aqueous lipid dispersion for inhalation via nebulization.
  * Administration procedures, volume and administration time are the same as for Arikace™.
  * Placebo will be administered for 28 days.
  Arms: Placebo

SUMMARY:
A major factor in the respiratory health of Cystic Fibrosis (CF) subjects is the prevalence of chronic Pseudomonas aeruginosa infections. The Pseudomonas aeruginosa infection rate in CF patients increases with age and by age 18 years approximately 85% of CF patients in the US are infected. Liposomal amikacin for inhalation (Arikace™) was developed as a possible treatment for chronic infection due to Pseudomonas aeruginosa in CF patients.

The purpose of this double-blind, placebo controlled study is to determine whether Arikace™ is effective in treating chronic lung infections caused by Pseudomonas aeruginosa in Cystic Fibrosis subjects. The study will enroll approximately 300 subjects in clinics in the US, Canada, Europe, Australia and New Zealand. Subjects will be randomized to 590 mg Arikace™ or placebo and will receive treatment for 28 days followed by a 56 day safety follow-up period. The subjects will be required to visit the clinic 8 times (including the Screening visit) over a period of approximately 3 months. No overnight stays at the clinic will be required. At the completion of the TR02-109 protocol, subjects who have consented and meet study safety criteria may enroll in the long-term, open-label, multi-cycle extension study of 590 mg of Arikace™ (under a separate protocol TR02-110).

DETAILED DESCRIPTION:
Cystic Fibrosis (CF) is a genetic disease resulting from mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene. Patients with CF manifest pathological changes in a variety of organs that express CFTR. The lungs are frequently affected often resulting in chronic infections by bacteria such as Pseudomonas aeruginosa and airway inflammation. Treatment of chronic lung infections is one of the principal goals of CF therapy. Arikace™ (liposomal amikacin for inhalation) is a sustained-release formulation of amikacin encapsulated inside nanoscale liposomal carriers designed for administration via inhalation. It is hypothesized that the sustained-release pulmonary targeting and biofilm penetration properties of this formulation will have several advantages over current therapies in treating CF patients with chronic lung infection caused by Pseudomonas aeruginosa.

This double blind, placebo controlled Phase 3 study has been designed to evaluate the efficacy, safety and tolerability of Arikace™ in treating CF patients with chronic bronchopulmonary infection. Eligible subjects will be randomized 1:1 to receive 590 mg of Arikace™ or placebo once daily using a PARI Investigational eFlow® Nebulizer. Subjects will receive 28 days of treatment and will then be followed for safety for 56 days. Total study duration is up to 102 days (~3 months) including an up to 18 day Screening period. Subjects will be evaluated for safety, tolerability and efficacy bi-weekly throughout the study. Pharmacokinetics (PK) of Arikace™ in blood, sputum and 24-hour urine will be determined in a subgroup of study subjects who consent to PK evaluation.

At the completion of the TR02-109 protocol, subjects who have consented and meet study safety criteria may enroll in the long-term, open-label, multi-cycle extension study of 590 mg of Arikace™ (under a separate protocol TR02-110).

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent or assent
* Confirmed diagnosis of CF
* History of chronic infection with Pseudomonas aeruginosa
* History of documented pulmonary exacerbation requiring treatment with antibiotics in the 12 months prior to Screening
* Sputum culture positive for Pseudomonas aeruginosa at Screening
* FEV1 ≥ 25% of predicted value at Screening

Key Exclusion Criteria:

* FEV1 <25% of predicted value at Screening
* History of hypersensitivity to aminoglycosides
* History of major complications of lung disease (including atelectasis, pneumothorax, major pleural effusion) within 8 weeks prior to Screening
* Hemoptysis of ≥60 mL in a 24-hour period within 4 weeks prior to Screening
* History of pulmonary tuberculosis or non-tuberculous mycobacterial lung disease treated within 2 years prior to Screening or requiring treatment at the time of Screening
* History of Allergic Broncho-Pulmonary Aspergillosis requiring systemic steroid treatment or any other condition requiring systemic steroids at a dose ≥ equivalent of 10 mg/day of prednisone within 3 months prior to Screening
* Presence of any clinically significant cardiac disease
* Active pulmonary malignancy (primary or metastatic) or any malignancy requiring chemotherapy or radiation therapy within one year prior to Screening or anticipated during the study period
* History of lung transplantation
* Daily, continuous oxygen supplementation or nighttime supplemental oxygen requirement of greater than 2 L/min
* Administration of any investigational products within 8 weeks prior to study Day 1
* Smoking tobacco or any substance within 6 months prior to Screening or anticipated inability to refrain from smoking throughout the study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Time to first protocol defined pulmonary exacerbation | 84 days

SECONDARY OUTCOMES:
Relative change in FEV1 (liters) and FEV1 (% predicted) | 84 days
Proportion of subjects experiencing protocol defined exacerbations | 84 days
Time to first antipseudomonal antibiotic treatment for pulmonary exacerbation | 84 days
Change in Pseudomonas aeruginosa and Burkholderia sp. density in sputum | 84 days
Change in patient reported outcomes/symptoms | 84 days
Evaluation of safety and tolerability | 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Gina Eagle, MD, Study Director — Insmed Incorporated